CLINICAL TRIAL: NCT06509984
Title: EBULO. a 20-Week Multicentre, Open Study Assessing the Efficacy and Safety of Apremilast in Patients > 6 Years of Age with EB Simplex Generalized
Brief Title: A 20-Week Study Assessing the Efficacy of Apremilast in Patients with EB Simplex Generalized
Acronym: EBULO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-PP-10; 2023-508794-83-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-15; First posted 2024-07-19 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Epidermolysis Bullosa Simplex; Genodermatosis
Keywords: Apremilast; Children; Pediatric
MeSH Terms: conditions — Epidermolysis Bullosa Simplex; Skin Diseases, Genetic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- apremilast treatment (Experimental): treatment by apremilast in two phases of challenge
  Interventions: Drug: Apremilast treatment

INTERVENTIONS:
Drug: Apremilast treatment — treatment of apremilast

SUMMARY:
The goal of this clinical trial is to Assessing the Efficacy and Safety of Apremilast in Patients > 6 years of age with EB simplex generalized . The main question it aims to answer are: describe efficacity of this treatment.

Participants will take treatments and have to use bullets during the study period.

DETAILED DESCRIPTION:
The patient will have 7 visits. After Confirmation of inclusion criteria and no exclusion criteria, the study will be explain to the patient after signing the inform consent and be included in the study Treatment Period (Period 1); challenge period This period will be the first treatment period that will occur from 8 weeks. During this period the patient will see the doctor at the hospital, he will perform the study procedures The second period : dechallenge (period 2): All patients stop their treatment for 4 weeks.

The second treatment period - rechallenge (period 3) the patient will take the treatment for a second 8 weeks period At week 20 - End of study

At each visit:

The investigator at each visit compliance to the treatment and adverse events, Measure vital signs and perform clinical examination.

The patient will assess the different questionnaires, for the study

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 6 years or older
* Laboratory confirmed diagnosis of EBS-sev due to KRT5 or 14 mutation (autosomal)
* Mean daily number of new blisters >3.
* Subject/caregiver agrees not to use any topical therapies other than the investigator approved

Exclusion Criteria:

* - EBS lesions requiring oral therapy to treat an infection
* Use of any diacerein containing product within 6 months prior to Visit 1
* Use of systemic immunotherapy or cytotoxic chemotherapy within 60 days prior to Visit 1
* Use of systemic steroidal therapy within 30 days prior to Visit 1
* Use of any systemic product that, in the opinion of the investigator, might put the subject at undue risk by study participation or interferes with the study assessments within 30 days prior to Visit 1

Ages: 6 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-06 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
To describe efficacy of apremilast | weeks 20
  number of new blister conting every day

SECONDARY OUTCOMES:
Safety of apremilast treatment | weeks 20
  number of SAE

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - CHU de Nice, Nice, France
  - APHP Necker-Enfants-Malades, Paris, France
  - APHP Hôpital Saint-Louis, Paris, France
  - chu de Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fontas E, Hubiche T, Maruani A, Moschoi R, Hussain S, Chiaverini C. Multicentre phase II open study assessing the efficacy and safety of apremilast in children and adults with epidermolysis bullosa simplex generalised: study protocol for the EBULO study. BMJ Open. 2025 Nov 12;15(11):e103194. doi: 10.1136/bmjopen-2025-103194. PMID 41224305